CLINICAL TRIAL: NCT05951920
Title: Lymph Node Aspiration to Decipher the Immune Response of Beta-variant Recombinant Protein Booster Vaccine (VidPrevtyn Beta, Sanofi) Compared to a Bivalent mRNA Vaccine (Comirnaty Original/Omicron BA.4-5, BioNTech-Pfizer) in Adults Previously Vaccinated With at Least 3 Doses of COVID-19 mRNA Vaccine. Ancillary of COVIBOOST 2
Brief Title: Lymph Node Aspiration to Decipher the Immune Response of Beta-variant Recombinant Protein Booster Vaccine (VidPrevtyn Beta, Sanofi) Compared to a Bivalent mRNA Vaccine (Comirnaty Original/Omicron BA.4-5, BioNTech-Pfizer) in Adults Previously Vaccinated With at Least 3 Doses of COVID-19 mRNA Vaccine.
Acronym: LymphoBOOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP230684; 2023-A01335-40 (Other: IDRCB ANSM)
Record Dates: First submitted 2023-07-06; First posted 2023-07-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: COVID-19
Keywords: COVID 19; mRNA vaccines; Immunology; Sub-unit vaccine; Booster; lymph nod; memory B cell
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymph node aspiration / Blood sampling (Experimental)
  Interventions: Procedure: Lymph node aspiration / Blood sampling

INTERVENTIONS:
Procedure: Lymph node aspiration / Blood sampling — Lymph node aspiration / Blood sampling

SUMMARY:
In order to investigate whether a germinal center response occurs following vaccine boost and to characterize it based on the type of vaccine received, we aim to analyze Spike and/or RBD-specific germinal center B cells within the draining lymph nodes.

To achieve this, we will perform lymph node fine needle aspiration of the draining lymph node in 6 subjects in each study arm, 3 to 6 weeks after the booster vaccine injection.

DETAILED DESCRIPTION:
Lymph nodes are secondary lymphoid organs essential for the establishment of the germinal center reaction, allowing the generation of long-lived B cell memory and high-affinity antibodies. In order to investigate whether a germinal center response occurs following vaccine boost and to characterize it based on the type of vaccine received, we aim to analyze Spike and/or RBD-specific germinal center B cells within the draining lymph nodes. Accessing germinal center through fine needle aspirations under ultrasound guidance has recently emerged as an innovative strategy in the United States to investigate vaccine response. This procedure under local anesthesia is well-tolerated, and no major side effects have been reported in a hundred patients who underwent fine needle aspiration. The technical details for performing this examination are now well-described.

Our previous work has highlighted the importance of repertoire diversity in responding to new variants of SARS-CoV-2. We thus aim to investigate whether a booster dose with mRNA or protein-based vaccine mobilizes memory B cells or naive cells, thereby contributing to a greater diversity of the Memory B cell comportment. To preserve the diversity of the memory B cell pool is absolutely essential for our immune system to adapt against variants.

To achieve this, we will perform lymph node fine needle aspiration of the draining lymph node in 6 subjects in each study arm, 3 to 6 weeks after the booster vaccine injection. Indeed, it has been shown that the response of germinal centers in response to a booster vaccination was detectable at 2- and 8-weeks post-injection vaccination.

This outpatient procedure will be performed by a radiologist under ultrasound guidance, aiming to collect 4 fine needle aspirations from 4 axillary draining lymph nodes under local anesthesia. Concurrently, a 35 mL blood sample will be collected from the subject to correlate the response in secondary lymphoid organs with the circulating response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and over included in COVIBOOST 2

Exclusion Criteria:

* Hypersensitivity to lidocaine, to anaesthetics of the amide type or to any of the excipients
* Patient with recurrent porphyrias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
The Spike and/or RBD-specific germinal center B cell response | Day 1
  As part of an ancillary study of COVIBOOST2 to analyse the percentage of Hu-1, Delta or Omicron Spike and RBD-specific germinal center B cells in draining lymph nodes 3-8 weeks after the Beta-variant recombinant protein booster vaccine (VidPrevtyn®Beta, Sanofi) or the bivalent mRNA vaccine (Comirnaty Original/Omicron BA.4-5, BioNTech-Pfizer), in adults previously vaccinated with at least 3 doses of COVID-19 mRNA vaccine, the last dose received at least 6 months prior the inclusion in the study.
The Spike and/or RBD-specific germinal center B cell repertoire | Day 1
  As part of an ancillary study of COVIBOOST2 to analyse the percentage of Hu-1, Delta or Omicron Spike and RBD-specific germinal center B cells in draining lymph nodes 3-8 weeks after the Beta-variant recombinant protein booster vaccine (VidPrevtyn®Beta, Sanofi) or the bivalent mRNA vaccine (Comirnaty Original/Omicron BA.4-5, BioNTech-Pfizer), in adults previously vaccinated with at least 3 doses of COVID-19 mRNA vaccine, the last dose received at least 6 months prior the inclusion in the study.

SECONDARY OUTCOMES:
The repertoire of the cellular germinal center B immune response in the two arms. | Day 1
  To determine the number of somatic hypermutations in the immunoglobulin heavy chain of each single Hu-1, Delta or Omicron Spike/RBD-specific germinal center cells. To determine the number of clonal relationships between Spike/RBD- specific germinal center B cells in draining lymph nodes with memory B cells in peripheral blood.

CONTACTS AND LOCATIONS:
Locations (1):
- GH Broca-Cochin-Hôtel-Dieu CIC 1417 Cochin-Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: No
The IPD will not be share. The 2 vaccines used in this study are marketed vaccine and used in routine care